CLINICAL TRIAL: NCT03827161
Title: GLANCE 2 - Glucosamine and Chondroitin (G&C) Effects Study
Brief Title: Glucosamine and Chondroitin in Preventing Inflammation in Overweight Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: RG1001578; NCI-2018-02647 (Other: CTRP)
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Healthy Subject; Overweight
MeSH Terms: conditions — Overweight | interventions — Glucosamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm I (glucosamine sulfate/chondroitin sulfate tablet) (Experimental): Patients receive glucosamine sulfate/chondroitin sulfate tablet PO on days 1-14 in the absence of disease progression or unacceptable toxicity. Fourteen days later, patients crossover to Arm II.
  Interventions: Dietary Supplement: Glucosamine
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO on days 1-14 in the absence of disease progression or unacceptable toxicity. Fourteen days later, patients crossover to Arm I.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Glucosamine — Given PO
  Arms: Arm I (glucosamine sulfate/chondroitin sulfate tablet)
Other: Placebo — Given PO
  Other Names: PLCB
  Arms: Arm II (placebo)

SUMMARY:
This trial studies glucosamine and chondroitin in preventing inflammation in overweight patients. Chronic inflammation contributes to cancer formation, and biomarkers of inflammation have been associated with cancer risk. Glucosamine and chondroitin may prevent inflammation and this trial may help identify the bacteria that help process them in the gut.

ELIGIBILITY:
Inclusion Criteria:

-Individuals from the Greater Seattle area who are overweight (body mass index [BMI] of 25-32.5 kg/m^2)

Exclusion Criteria:

* Chronic medical illness, history of gastrointestinal, hepatic, or renal disorders, or inflammatory conditions (including autoimmune and inflammatory diseases)
* Pregnancy or lactation
* Currently on a weight-loss diet
* BMI (body mass index) < 25 or > 32.5 kg/m^2
* Alcohol intake of greater than 2 drinks/day (2 drinks being equivalent to 720 ml beer, 240 ml wine or 90 ml spirits)
* Current use of prescription or over-the-counter medications other than oral contraceptives and hormone secreting intrauterine device (IUD)s, multivitamin pills or infrequent use of aspirin and nonsteroidal anti-inflammatory drugs (NSAIDs), or use of aspirin or NSAIDs more than 2 days per week
* Abnormal renal, liver or metabolic test
* Inability to swallow pills
* Known allergy to shellfish
* Not willing to take pills made from shellfish or animal sources
* Intention to relocate out of study area within next 2 months
* Any antibiotic use in the past 6 months

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Effects of glucosamine sulfate/chondroitin sulfate tablet (G&C) on gut microbial community modulation | Up to 2 years
  shifts in the bacterial communities within person based on clustering of operational taxonomic units (OTU) at 97% utilizing principal coordinate analysis [PCOA]).
Effects of G&C on serum C-reactive protein (CRP) | Up to 2 years
  evaluated using a generalized estimating equation which accounts for variation due to repeated measures within an individual

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Lampe, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No